CLINICAL TRIAL: NCT06430463
Title: Effect of Interscalenous Block Anesthesia on Hearing Levels
Brief Title: Impact of Interscalenous Block Anesthesia on Hearing
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 02-2024/11
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-10

CONDITIONS: Hearing Loss
Keywords: hearing level; interscalene block anesthesia
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry, Speech; Acoustic Impedance Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing shoulder surgery with interscalene block: Ultrasound-guided Interscalene block will be applied to all patientsand also every patients will be treated with the same multimodal analgesia for postoperative pain control. The patient will be examined by ENT physician on the morning of the operation, after a detailed anamnesis. otoscopic examination will be performed, pure tone audiometry, speech audiometry and tympanometric examination will be performed and recorded.The same tests will be performed at the next day after the surgery but before the discharge and also when he/she applies for the first week check-up.
  Interventions: Diagnostic Test: pure tone audiometry levels

INTERVENTIONS:
Diagnostic Test: pure tone audiometry levels — The patient will be examined by ENT physician on the morning of the operation, otoscopic examination will be performed, pure tone audiometry, speech audiometry and tympanometric examination will be performed and recorded.The same tests will be performed at the next day after the surgery but before the discharge and also when he/she applies for the first week check-up.
  Other Names: speech audiometry; tympanometry; otoscopic examnation

SUMMARY:
Interscalene brachial plexus block (ISBPB) is used frequently in shoulder, clavicle and upper arm surgeries to obtain analgesia in the postoperative period. Our primary aim in this study is to evaluate if interscalene block anesthesia has an effect on hearing levels of patients undergoing orthopedic shoulder surgeries.

DETAILED DESCRIPTION:
Interscalene brachial plexus block (ISBPB) is used for both anesthesia and analgesia purposes in shoulder, clavicle and upper arm surgeries. It is also frequently used to obtain analgesia in the postoperative period especially in patients undergoing shoulder surgeries. Thus, it provides decrease in opioid need and opioid related side effects in the perioperative period. The effect of IBPB on hearing is probably not caused by an effect on the vestibulocochlear nerve because of its central location. The innervation area of the greater auricular nerve, a derivative of the cervical plexus, is often involved in an IBPB. However, this nerve is not known to affect hearing. The nerves supplying the outer ear canal and the tympanic membrane (branches of the mandibular, facial and vagal nerves) are located far enough from the IBPB injection site to make their involvement unlikely. However, sound conduction through the middle ear to the inner ear, and functioning of the spiral organ of the cochlea may be indirectly affected by regional sympathetic block that is most likely seen after IBPB. Sympathetic block may cause vasodilatation and swelling of the mucosal membranes of the middle ear and the eustachian tube with deterioration of hearing.

The patient will be examined by ENT physician on the morning of the operation, after a detailed anamnesis. otoscopic examination will be performed, pure tone audiometry, speech audiometry and tympanometric examination will be performed and recorded.The same tests will be performed at the next day after the surgery but before the discharge and also when he/she applies for the first week check-up. Ultrasaoun guided Interscalene block anesthesia will be applied to all patients. Each patient will be treated with the same multimodal analgesia method at the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* participants are undergoing a shoulder surgery.
* ASA I and II patients without uncontrolled diabetes and hypertension
* participants have normal or near-normal hearing thresholds in the un-operated ear

Exclusion Criteria:

* participants have hearing loss (PTA > 35 dB HL) in pure tone audiometry testing before surgery in any side
* participants have medical conditions after the surgery which prevents having hearing tests
* participants have abnormal tympanometric results
* participants with chronic otitis media or a history of ear surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing shoulder surgery with ultrasoun-guided interscalene brachial plexus block.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Difference of 10 dB or more between Pre- and Post-surgery pure tone audiometry measurements at any Frequency | pre-surgery, a day after surgery
  pure tone audiometry measurements at all frequencies measured via MADSEN Astera2 device

CONTACTS AND LOCATIONS:
Locations (1):
- Karaman training and research hospital, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided